CLINICAL TRIAL: NCT05814900
Title: Investigation of Mohs Surgical Margins Using Two Photon Microscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Rochester Dermatologic Surgery (Other)
Responsible Party: Principal Investigator, Michael Giacomelli, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00008153
Record Dates: First submitted 2023-03-31; First posted 2023-04-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-07

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TPFM imaging of surgical margins (Experimental): Patients will be imaged with TPFM
  Interventions: Device: Two photon microscopy imaging

INTERVENTIONS:
Device: Two photon microscopy imaging — Excised tissues will be imaged with two photon microscopy

SUMMARY:
The goal of this clinical trial is to compare the use of two photon fluorescence microscopy for detecting residual basal cell carcinoma during Mohs surgery. The main question it aims to answer is:

• How similar are diagnosis of surgical margins to on two photon fluorescence microscopy compared to frozen section histology

DETAILED DESCRIPTION:
This study is an study of skin cancer that will evaluate the feasibility of two photon fluorescence microscopy (TPFM) to evaluate surgical margins followed by standard of care frozen section analysis (FSA) for confirmation. To protect patients, following TPFM imaging, patients will receive standard of care evaluation using cryosectioned H&E slides, thus all patients will receive standard of care confirmation following experimental imaging.

Individual excisions from consenting patients will be selected, fluorescently labeled and diagnosed using TPFM. Following imaging, specimens will be cryosectioned as per normal procedure. Following treatment, the results of the TPFM evaluation of each Mohs excisions will be compared to the results from FSA to assess the overall accuracy of TPFM and to determine if TPFM would result in changes to patient care if used without FSA confirmation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing treatment for BCC with Mohs surgery at the performance site
* Able to read and understand consent form

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Agreement between frozen sections and two photon microscopy on Mohs margins | During Mohs surgery
  The fraction of Mohs surgical margins in which TPFM agrees with FSA will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Giacomelli, Ph.D, Principal Investigator — University of Rochester
Locations (1):
- Rochester Dermatologic Surgery, Victor, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ching-Roa VD, Huang CZ, Ibrahim SF, Smoller BR, Giacomelli MG. Real-time Analysis of Skin Biopsy Specimens With 2-Photon Fluorescence Microscopy. JAMA Dermatol. 2022 Oct 1;158(10):1175-1182. doi: 10.1001/jamadermatol.2022.3628. PMID 36069886